CLINICAL TRIAL: NCT07347418
Title: Phase 1, Open Label, Dose Escalation Study to Evaluate the Safety, Expansion, Persistence, and Preliminary Clinical Activity of Autologous CD64 CAR T Cells in Patients With Relapsed and/or Refractory Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (HR-MDS)
Brief Title: CD64 CAR T Cell Therapy in Adults With Relapsed and/or Refractory AML or HR-MDS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0718.cc
Record Dates: First submitted 2025-12-01; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Refractory Acute Myeloid Leukemia (AML); High-risk Myelodysplastic Syndrome (MDS); Relapsed Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)/AML; Myelodysplastic Syndrome; AML (Acute Myeloid Leukemia)
Keywords: AML; MDS; CD64; CAR T; CAR T cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: All participants receive CD64 CAR T cells. There is no control arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relapsed and/or Refractory AML and HR-MDS (Experimental): Patients with relapsed and/or refractory acute myeloid leukemia (AML) or high-risk myelodysplastic syndromes (HR-MDS) will receive lymphodepleting chemotherapy followed by infusion of CD64 CAR T-cells, starting at dose level 1.
  Interventions: Drug: CD64 CAR T Cells

INTERVENTIONS:
Drug: CD64 CAR T Cells — CD64 CAR T is a lentiviral transduced autologous T cells expressing anti-CD64 chimeric antigen receptors (CAR) possessing tandem CD3ζ and 4-1BB (CD3ζ/4-1BB) costimulatory domains.

SUMMARY:
This is a Phase 1, open label, dose-escalation study to evaluate the safety, expansion, persistence, and preliminary clinical activity of lentivirally transduced autologous T cells expressing anti-CD64 chimeric antigen receptors (CAR) expressing tandem CD3ζ and 4-1BB (CD3ζ/4-1BB) costimulatory domains in subjects with refractory or relapsed (R/R) acute myeloid leukemia (AML) or high-risk myelodysplastic syndromes (MDS). This CAR T cell product will be referred to as "CD64 CAR T" which is CD64 directed, autologous, genetically modified CAR T cells. The primary objective identify the safety profile and maximum tolerated dose (MTD) of CD64 CAR T in subjects with R/R AML or MDS as determined by the defined DLTs using a standard Bayesian Optimal Interval (BOIN) design.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Subjects must have one of the following diagnoses per the International Consensus Classification (ICC) 2022 criteria:

   1. Acute Myeloid Leukemia (AML).
   2. Myelodysplastic Syndrome/Acute Myeloid Leukemia (MDS/AML).
   3. MDS with excess blasts (MDS-EB).
3. Refractory OR relapsed AML, MDS/AML, or MDS-EB, defined as:

   a. Refractory disease i. Lack of at least PR after a minimum of 1 cycle of a hypomethylating agent (HMA) and venetoclax (Ven) combination (Ven/HMA) OR; ii. Lack of CRMRD- after a minimum of 3 cycles of Ven/HMA (MRD defined as ≥ 0.1% blasts by multi-parameter flow cytometry).

   b. Relapsed disease i. Recurrence of > 5% blasts in the bone marrow by morphology OR; ii. ≥ 0.1% blasts by multi-parameter flow cytometry when a previous bone marrow aspirate demonstrated MRD-negativity OR; iii. ≥ 0.1% blasts by multi-parameter flow cytometry ≥ 6 months post-allogeneic stem cell transplant AND no active graft-versus-host disease (GVHD) requiring immunosuppressive therapy.
4. Subjects must have received at least one prior line of therapy, including at least one line of therapy containing Ven.
5. Documentation of CD64 expression on myeloid blasts by flow cytometry after the most recent relapse, as determined by standardized and validated multiparameter flow cytometry assay (Hematologics, Inc., Seattle, WA).
6. Total white blood cell (WBC) count ≤ 25 x 109/L prior to apheresis. Hydroxyurea is permitted to achieve this.
7. Absolute lymphocyte count (ALC) ≥ 200/µL prior to apheresis OR ALC < 200 µL with concurrent lymphocyte subset analysis (CD3, CD4, and CD8 counts) confirming an absolute CD3 count ≥ 150/µL.
8. Confirmed availability of cells for a rescue stem cell transplant AND subject must be deemed an appropriate candidate for such therapy per institutional standards.
9. Subjects who have undergone prior allogeneic stem cell transplant must be ≥ 6 months out from transplant and be off systemic immunosuppression for at least 1 month at the time of enrollment.
10. Adequate organ function, defined as:

    1. Creatinine clearance ≥ 30 mL/min, based on the CKD-EPI Creatinine Equation (2021).
    2. AST/ALT ≤ 5x upper limit of the normal range, unless considered to be due to leukemic involvement.
    3. Bilirubin ≤ 3x upper limit of the normal range, unless the subject has Gilbert's Syndrome or considered to be due to leukemic involvement.
    4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air, unless considered to be due to leukemic involvement.
    5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA.
11. ECOG performance status 0, 1, or 2.
12. Signed informed consent form.
13. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in the protocol main text.
14. Willing to participate in the long-term follow-up protocol that is required if CAR T cell therapy is administered.

Exclusion Criteria:

1. Subjects with Acute Promyelocytic Leukemia (APL) with t(15;17)
2. Receipt of previous chemotherapy for AML or MDS, as follows:

   a. Prior to apheresis, the following washout periods apply: i. Hydroxyurea: 1 day ii. Hypomethylating agent and/or venetoclax: 7 days iii. Small molecule targeted therapy (including tyrosine kinase inhibitors): 3 half-lives or 7 days, whichever is shorter.

   iv. Immune checkpoint inhibitors or other immunological agents: 5 half-lives or 28 days, whichever is shorter.

   v. Investigational products: 5 half-lives or 28 days, whichever is shorter. vi. Any other systemic chemotherapy: 14 days vii. Allogeneic stem cell transplantation: 180 days viii. Donor lymphocyte infusion (DLI): 60 days ix. Craniospinal or total body radiation: 42 days b. After apheresis and prior to lymphodepletion, no treatment for AML and MDS is permitted, with the exception of bridging hydroxyurea with a washout period of 1 day prior to the start of the lymphodepletion regimen.
3. Concurrent use of systemic steroids or immunosuppressant medications. Recent or current use of inhaled steroids or physiologic replacement with hydrocortisone is not exclusionary.
4. Previous treatment with investigational gene or cell therapy (including CAR therapy).
5. Signs or symptoms indicative of CNS leukemia involvement. A CNS evaluation should be performed if CNS involvement is suspected to rule out CNS leukemia involvement.
6. Pregnant or lactating (nursing) women.
7. Known HIV infection or active Hepatitis B or Hepatitis C infection.
8. Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
9. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
10. Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to leukemia or previous leukemia treatment.
11. Subjects with cardiac arrhythmia, or arrhythmias that are not stable with medical management, within 2 weeks of the Screening/Enrollment visit.
12. Any uncontrolled active medical disorder that would preclude participation as outlined.
13. Evidence of another uncontrolled malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Day 0 through Day 42
  MTD will be established from the DLTs, which will be considered from the time of CD64 CAR T infusion (Day 0) through Day 42 after the subject's last infusion. A DLT is a treatment-emergent adverse event, or a clinically significant abnormal laboratory value, observed during the DLT observation period.

SECONDARY OUTCOMES:
Manufacturability - Product Release Failure | Day 0 (Infusion)
  The proportion of CD64 CAR T products that fail to meet the product release criteria, out of the number of enrolled subjects in whom manufacturing was attempted.
Manufacturability - Dose Failures | Day 0 (Infusion)
  The proportion of CD64 CAR T products that fail to meet the assigned dose, out of the number of subjects enrolled for whom manufacturing was attempted.
Efficacy - Overall Response Rate (ORR) | Day 28, Month 3, and Month 6
  The efficacy of the CD64 CAR T-cell product will be assessed by determining the overall response rate (ORR) through morphologic evaluation of bone marrow at Day 28 post-infusion. Response categories include complete remission (CR), CR with measurable residual disease negative (CR MRD-), CR with incomplete hematologic recovery (CRi), CR with partial hematologic recovery (CRh), morphological leukemia-free state (MLFS), and partial response (PR).
Efficacy - Overall Survival | Up to 12 months post infusion
  Overall Survival (OS) will be measured from date of CD64 CAR T-cell infusion until death from any cause. At one year post-infusion, OS will be analyzed using Kaplan-Meier estimates.
Efficacy - Progression Free Survival (PFS) | From treatment to end of study
  Progression free survival (PFS) is defined as the time from CD64 CAR T cell infusion to the time of disease progression or death from any cause. Disease progression will be determined based on morphologic assessment of bone marrow and other relevant clinical criteria. Subjects who withdraw consent during the study, lost to follow-up, or complete follow-up with no events will be censored.
Efficacy - Duration of Response (DOR) | From treatment to end of study
  Duration of Response (DoR) will be evaluated with the Kaplan-Meier responses for subjects who achieve CR, CRMRD- (measurable residual disease negative), CRi, CRh, MLFS (morphological leukemia-free state), and partial response (PR) using on-study assessments.
Efficacy - Need for Rescue Allogenic Stem Cell Transplant | From treatment to early termination for transplant
  The proportion of subjects who require a rescue allogenic stem cell transplant following CD64 CAR T-cell infusion due to lack of response, disease progression, or relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Angelos, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States